CLINICAL TRIAL: NCT02558894
Title: A Phase II Open-Label, Multi-Center Study of MEDI4736 Evaluated as Single Agent or in Combination With Tremelimumab in Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Phase II Study of MEDI4736 Monotherapy or in Combinations With Tremelimumab in Metastatic Pancreatic Ductal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4198C00001
Record Dates: First submitted 2015-08-27; First posted 2015-09-24 (Estimated); Results first posted 2018-08-02 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Ductal Adenocarcinoma, PDAC
MeSH Terms: conditions — Anophthalmia with pulmonary hypoplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MEDI4736 monotherapy (Experimental): MEDI4736 via IV infusion.
  Interventions: Drug: MEDI4736 monotherapy
- tremelimumab+MEDI4736 (Experimental): MEDI4736+tremelimumab via IV infusion.
  Interventions: Drug: tremelimumab+MEDI4736

INTERVENTIONS:
Drug: MEDI4736 monotherapy — MEDI4736 via IV infusion.
  Arms: MEDI4736 monotherapy
Drug: tremelimumab+MEDI4736 — tremelimumab+MEDI4736 via IV infusion.
  Arms: tremelimumab+MEDI4736

SUMMARY:
A Phase II Open-Label, Multi-Center Study of MEDI4736 Evaluated as Single Agent or in Combination with Tremelimumab in Patients with Metastatic Pancreatic Ductal Adenocarcinoma.

DETAILED DESCRIPTION:
This is a Phase II, open-label, multi-center study to determine the efficacy and safety of MEDI4736 evaluated as single agent or in combination with tremelimumab in patients with metastatic pancreatic ductal adenocarcinoma (PDAC) whose disease has progressed on fluoropyrimidine containing or gemcitabine-containing first-line chemotherapy.This study will consist of Part A, lead-in, as well as a possible expansion Part B.

ELIGIBILITY:
Inclusion Criteria: -

1. Histologically or cytologically confirmed metastatic PDAC, no more than 1 prior chemotherapy regimen
2. Eastern Cooperative Oncology Group 0 or 1
3. At least 1 lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) scan and that is suitable for accurate repeated measurements

Exclusion Criteria:

1. Any concurrent chemotherapy, investigational product , biologic, or hormonal therapy for cancer treatment.
2. History of leptomeningeal carcinomatosis
3. Ascites requiring intervention
4. Brain metastases or spinal cord compression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-11-16 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen M O'Reilly, M.D, Principal Investigator — Memorial Sloan Kettering Cancer Center, 300 East 66th Street,New York,NY 10065
Locations (17):
- United States (2):
  - Research Site, Tampa, Florida
  - Research Site, New York, New York
- Canada (5):
  - Research Site, Vancouver, British Columbia
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Germany (3):
  - Research Site, Friedrichshafen
  - Research Site, München
  - Research Site, Tübingen
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Groningen
  - Research Site, Nijmegen
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (2):
  - Research Site, Barcelona
  - Research Site, Madrid

REFERENCES:
- [Derived] O'Reilly EM, Oh DY, Dhani N, Renouf DJ, Lee MA, Sun W, Fisher G, Hezel A, Chang SC, Vlahovic G, Takahashi O, Yang Y, Fitts D, Philip PA. Durvalumab With or Without Tremelimumab for Patients With Metastatic Pancreatic Ductal Adenocarcinoma: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2019 Oct 1;5(10):1431-1438. doi: 10.1001/jamaoncol.2019.1588. PMID 31318392
- See also: redacted csp — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3297&filename=d4198c00001-revised-csp-002973340_CORRECT-redact.pdf
- See also: Redacted SAP — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3297&filename=d4198c00001-statistical-analysis-plan-edition-2_ID-003081403-redact.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 16 Nov 2015; Part A data cut-off: 26 May 2017. The study contained a Part B which was not opened; only Part A was conducted.
  Study assessed efficacy of durvalumab (MEDI4736) + tremelimumab combination therapy compared to durvalumab (MEDI4736) monotherapy.
  Study performed at 21 sites in 6 countries.
Pre-assignment Details: 65 patients were randomised to receive investigational product (IP) and 64 received treatment. One randomised patient in the durvalumab monotherapy arm was withdrawn prior to receiving any IP but was still included in the full analysis set (FAS) which was used for participant flow and baseline analysis.
Groups:
- Durvalumab (MEDI4736) Plus Tremelimumab: Patients in the durvalumab (MEDI4736) plus tremelimumab combination therapy arm received 1.5 grams (g) durvalumab and 75 milligrams (mg) tremelimumab via intravenous (IV) infusion every 4 weeks (q4w) over a 16-week treatment period. Patients then continued with durvalumab monotherapy at 1.5 g q4w, beginning at Week 16, 4 weeks after the last dose of combination therapy, up to a total of 9 additional doses, with the final dose at Week 48.
  For the combination therapy, tremelimumab was administered first; the durvalumab infusion was started approximately 1 hour after the end of the tremelimumab infusion.
- Durvalumab (MEDI4736) Monotherapy: Patients in the durvalumab (MEDI4736) monotherapy arm received 1.5 g durvalumab via IV infusion q4w over a 48-week treatment period (up to 13 doses).
Period: Overall Study
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab | Durvalumab (MEDI4736) Monotherapy
Started | 32 | 33
Patients Who Received IP | 32 | 32
Completed | 0 | 0
Not Completed | 32 | 33
Not completed — Death; any cause, entire study duration | 28 | 31
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Closure of Part A | 2 | 1

BASELINE CHARACTERISTICS:
Population: All patients in the FAS who were randomised to treatment were included in the baseline analysis.
Groups:
- Durvalumab (MEDI4736) Plus Tremelimumab: Patients in the durvalumab (MEDI4736) plus tremelimumab combination therapy arm received 1.5 g durvalumab and 75 mg tremelimumab via IV infusion q4w over a 16-week treatment period. Patients then continued with durvalumab monotherapy at 1.5 g q4w, beginning at Week 16, 4 weeks after the last dose of combination therapy, up to a total of 9 additional doses, with the final dose at Week 48.
  For the combination therapy, tremelimumab was administered first; the durvalumab infusion was started approximately 1 hour after the end of the tremelimumab infusion.
- Total: Total of all reporting groups
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab | Durvalumab (MEDI4736) Monotherapy | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (9.60) | 61.6 (9.54) | 61.5 (9.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 31
  Male | 15 | 19 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 30 | 33 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 10 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 17 | 22 | 39
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) in All Patients Using Investigator Assessments According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: ORR was defined as the percentage of patients with at least one visit response of confirmed complete response (CR) or partial response (PR). CR was defined as disappearance of all target lesions (TLs) since baseline. Any pathological lymph nodes selected as TLs must have had reduction in short axis to <10 millimeters (mm). PR was defined as at least a 30% decrease in the sum of diameters of TLs, taking as reference the baseline sum of diameters. A confirmed response meant that a response of CR/PR was recorded at 1 visit and confirmed by repeat imaging, preferably at the next regularly scheduled imaging visit and not less than 4 weeks after the visit when response was first observed with no evidence of progression between the initial and CR/PR confirmation visits. Results are reported as percentage of patients with a confirmed response and percentage of patients with confirmed or unconfirmed responses (i.e., including single visit responses).
Time Frame: From date of first infusion until confirmed disease progression or death (up to approximately 18 months for the data analysis cut-off)
Population: The FAS included all randomised patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab | Durvalumab (MEDI4736) Monotherapy
Number analyzed (Participants) | 32 | 33
Percentage of participants
  Confirmed responses only | 3.1 [0.08 to 16.22] | 0 [0 to 10.58]
  Confirmed and unconfirmed responses | 3.1 [0.08 to 16.22] | 6.1 [0.74 to 20.23]

2. Secondary Outcome: Progression-free Survival (PFS) Using Investigator Assessments According to RECIST 1.1
Description: PFS was defined as the time from the date of randomisation until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient had withdrawn from randomised therapy or had received another anti-cancer therapy prior to progression. Results are reported as median time from randomisation to PFS, calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 1
Population: The FAS included all randomised patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab | Durvalumab (MEDI4736) Monotherapy
Number analyzed (Participants) | 32 | 33
Months | 1.5 [1.2 to 1.5] | 1.5 [1.3 to 1.5]

3. Secondary Outcome: PFS Rate at 3 Months and at 6 Months
Description: PFS was defined as the time from the date of randomisation until the date of objective disease progression or death (by any cause in the absence of progression) regardless of whether the patient had withdrawn from randomised therapy or had received another anti-cancer therapy prior to progression. PFS rates were calculated using Kaplan-Meier estimates of the cumulative probability of PFS. The PFS rate at 3 months and 6 months was equivalent to the percentage of patients with PFS after 3 months and 6 months, respectively.
Time Frame: From date of first infusion until confirmed disease progression or death (up to 3 months and 6 months)
Population: The FAS included all randomised patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab | Durvalumab (MEDI4736) Monotherapy
Number analyzed (Participants) | 32 | 33
Percentage of participants
  PFS rate at 3 months | 9.4 [2.4 to 22.3] | 10.9 [3.0 to 24.7]
  PFS rate at 6 months | 9.4 [2.4 to 22.3] | 3.6 [0.3 to 15.4]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomisation until death due to any cause. Results are reported as median OS, calculated using the Kaplan-Meier technique.
Time Frame: From date of first infusion until death (up to approximately 18 months for the data analysis cut-off)
Population: The FAS included all randomised patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab | Durvalumab (MEDI4736) Monotherapy
Number analyzed (Participants) | 32 | 33
Months | 3.1 [2.2 to 6.1] | 3.6 [2.7 to 6.1]

5. Secondary Outcome: Survival Status, Presented as OS Rate, at 6 Months and at 12 Months
Description: OS was defined as the time from the date of randomisation until death due to any cause. OS rates were calculated using Kaplan-Meier estimates of the cumulative probability of survival at each indicated time period. The OS rate at 6 months and 12 months was equivalent to the percentage of patients with OS after 6 months and 12 months, respectively.
Time Frame: From date of first infusion until death (up to 6 months and 12 months)
Population: The FAS included all randomised patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab | Durvalumab (MEDI4736) Monotherapy
Number analyzed (Participants) | 32 | 33
Percentage of participants
  Survival rate at 6 months | 36.2 [20.0 to 52.7] | 34.9 [19.2 to 51.1]
  Survival rate at 12 months | 8.8 [1.8 to 22.8] | 6.3 [1.1 to 18.4]

6. Secondary Outcome: Best Objective Response (BoR) Using Investigator Assessments According to RECIST 1.1
Description: BoR was calculated based on the overall visit responses from each RECIST assessment. It was the best response a patient had following date of first dosing but prior to starting any subsequent cancer therapy and prior to RECIST progression or last evaluable assessment in absence of RECIST progression. Categorisation of BoR was based on RECIST using the following response categories: CR and PR for status of 'Response'; Stable Disease (SD) ≥6 weeks, Progressive Disease (PD) and Not Evaluable (NE) for status of 'Non-response'. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. PD was defined as at least a 20% increase in the sum of diameters of TLs taking as reference the smallest sum on study. NE was only relevant if any of the TLs were not assessed or not evaluable or had a lesion intervention at this visit. Results are reported as number of patients with BoR for each of the indicated categories.
Time Frame: as for outcome 1
Population: The FAS included all randomised patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab | Durvalumab (MEDI4736) Monotherapy
Number analyzed (Participants) | 32 | 33
Participants
  Response: Total | 1 | 0
  Response: CR | 0 | 0
  Response: PR | 1 | 0
  Non-response: Total | 31 | 33
  Non-response: Stable disease ≥6 weeks | 5 | 7
  Non-response: Progression of disease | 26 | 25
  Non-response: Not evaluable | 0 | 1

7. Secondary Outcome: Disease Control Rate (DCR) Using Investigator Assessments According to RECIST 1.1
Description: DCR at 3 months was defined as the percentage of patients who have a BoR of CR or PR in the first 3 months or who have demonstrated SD for a minimum interval of 13 weeks following the start of treatment. DCR at 6 months was defined as the percentage of patients who have a BoR of CR or PR in the first 6 months or who have demonstrated SD for a minimum interval of 26 weeks following the start of treatment. DCR at 12 months was defined as the percentage of patients who have a BoR of CR or PR in the first 12 months or who have demonstrated SD for a minimum interval of 52 weeks following the start of treatment. Results are reported as the percentage of patients with disease control for each of the indicated categories.
Time Frame: From date of first infusion until confirmed disease progression or death (up to 3 months, 6 months and 12 months)
Population: The FAS included all randomised patients.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab | Durvalumab (MEDI4736) Monotherapy
Number analyzed (Participants) | 32 | 33
Percentage of participants
  At 3 months | 9.4 [1.98 to 25.02] | 6.1 [0.74 to 20.23]
  At 6 months | 6.3 [0.77 to 20.81] | 0 [0.00 to 10.58]
  At 12 months | 3.1 [0.08 to 16.22] | 0 [0.00 to 10.58]

8. Secondary Outcome: Pharmacokinetics (PK) of Durvalumab (MEDI4736)
Description: To evaluate PK, blood samples were collected pre- and post-dose and durvalumab (MEDI4736) concentrations in serum were determined. On Day 1 of Cycles 1, 4 and 7 (Weeks 0, 12 and 24), PK samples were collected pre-dose (within 60 minutes prior to treatment with any IP) and post-dose at the end of infusion (within 10 minutes of end of infusion of durvalumab and within 10 minutes of end of infusion of tremelimumab [for patients receiving durvalumab plus tremelimumab]). On Day 1 of Cycle 2 (Week 4), PK samples were collected pre-dose (within 60 minutes prior to treatment with any IP) only. The 3-month follow-up sample for durvalumab was relative to the respective last dose. Results are reported as mean pre- or post-dose durvalumab concentrations as indicated by the individual categories (1 cycle=4 weeks). Samples below lower limit of quantification were treated as missing in the analyses.
Time Frame: Blood samples were collected pre-dose on Day 1 (Week 0), Week 4, Week 12 and Week 24, post-dose on Day 1, Week 12 and Week 24, and additionally at 3 months after the last dose (follow-up).
Population: The PK analysis set included all patients who received at least 1 dose of IP, and had PK sampling data post-dose without important deviations or events to affect PK (n=64). Only patients with data available at the timepoints of testing were included in the analyses.
Measure: Mean (Standard Deviation); unit: Micrograms per millilitre (mcg/mL)
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab | Durvalumab (MEDI4736) Monotherapy
Number analyzed (Participants) | 32 | 32
Micrograms per millilitre (mcg/mL)
  Cycle 1, Day 1, pre-infusion (Day 1): number analyzed (Participants) | 3 | 0
  Cycle 1, Day 1, pre-infusion (Day 1) | 217.338 (345.4913) |
  Cycle 1, Day 1, post-infusion (Day 1): number analyzed (Participants) | 31 | 31
  Cycle 1, Day 1, post-infusion (Day 1) | 566.078 (151.4199) | 562.218 (152.3811)
  Cycle 2, Day 1, pre-infusion (Day 29): number analyzed (Participants) | 22 | 21
  Cycle 2, Day 1, pre-infusion (Day 29) | 100.417 (39.7229) | 98.668 (36.5072)
  Cycle 4, Day 1, pre-infusion (Day 85): number analyzed (Participants) | 6 | 6
  Cycle 4, Day 1, pre-infusion (Day 85) | 236.205 (98.8964) | 228.450 (36.8395)
  Cycle 4, Day 1, post-infusion (Day 85): number analyzed (Participants) | 5 | 6
  Cycle 4, Day 1, post-infusion (Day 85) | 825.818 (322.8247) | 760.456 (100.6974)
  Cycle 7, Day 1, pre-infusion (Day 169): number analyzed (Participants) | 3 | 1
  Cycle 7, Day 1, pre-infusion (Day 169) | 166.736 (47.3872) | 152.706 (NA) — Data applies to one patient so standard deviation value not applicable.
  Cycle 7, Day 1, post-infusion (Day169): number analyzed (Participants) | 3 | 1
  Cycle 7, Day 1, post-infusion (Day169) | 918.270 (98.4286) | 825.578 (NA) — Data applies to one patient so standard deviation value not applicable.
  3-month follow-up: number analyzed (Participants) | 1 | 4
  3-month follow-up | 38.456 (NA) — Data applies to one patient so standard deviation value not applicable. | 19.684 (20.2664)

9. Secondary Outcome: PK of Tremelimumab
Description: To evaluate PK, blood samples were collected pre- and post-dose and tremelimumab concentrations in serum were determined. On Day 1 of Cycles 1 and 4 (Weeks 0 and 12), PK samples were collected pre-dose (within 60 minutes prior to treatment with any IP) and post-dose at the end of infusion (within 10 minutes of end of infusion of tremelimumab). On Day 1 of Cycle 2 (Week 4), PK samples were collected pre-dose (within 60 minutes prior to treatment with any IP) only. The 3-month follow-up sample for tremelimumab was relative to the respective last dose. Results are reported as mean pre- or post-dose tremelimumab concentrations as indicated by the individual categories (1 cycle=4 weeks). Samples below lower limit of quantification were treated as missing in the analyses.
Time Frame: Blood samples were collected pre-dose on Day 1 (Week 0), Week 4 and Week 12, post-dose on Day 1 and Week 12, and additionally at 3 months after the last dose (follow-up).
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab
Number analyzed (Participants) | 32
mcg/mL
  Cycle 1, Day 1, pre-infusion (Day 1): number analyzed (Participants) | 2
  Cycle 1, Day 1, pre-infusion (Day 1) | 13.114 (11.7182)
  Cycle 1, Day 1, post-infusion (Day 1): number analyzed (Participants) | 30
  Cycle 1, Day 1, post-infusion (Day 1) | 24.477 (6.3516)
  Cycle 2, Day 1, pre-infusion (Day 29): number analyzed (Participants) | 23
  Cycle 2, Day 1, pre-infusion (Day 29) | 4.880 (2.2623)
  Cycle 4, Day 1, pre-infusion (Day 85): number analyzed (Participants) | 6
  Cycle 4, Day 1, pre-infusion (Day 85) | 8.753 (4.9962)
  Cycle 4, Day 1, post-infusion (Day 85): number analyzed (Participants) | 6
  Cycle 4, Day 1, post-infusion (Day 85) | 21.150 (5.8997)
  3-month follow-up: number analyzed (Participants) | 0

10. Secondary Outcome: Presence of Antidrug Antibodies (ADAs) for Durvalumab (MEDI4736)
Description: ADA prevalence was the proportion of the ADA evaluable set who had an ADA positive result at any point in time, baseline or post-baseline. ADA incidence (treatment-emergent ADA) was the sum of both treatment-induced (post-baseline ADA positive only) and treatment-boosted ADA positive patients as a proportion of the evaluable patient population. Treatment-boosted ADA was defined as baseline positive ADA titre boosted to a 4-fold or higher level following IP administration. Persistently positive was defined as positive at ≥2 post-baseline assessments (with ≥16 weeks between first and last positive) or positive at last post-baseline assessment. Transiently positive was defined as at least 1 post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive. Results are reported as number of patients with detectable anti-durvalumab antibodies satisfying each of the indicated categories. Note: 'positive' is denoted by 'pos' in some category titles.
Time Frame: Immunogenicity samples were collected on Day 1 (Week 0), Week 4, Week 12 and Week 24, and additionally at 3 months and 6 months after the last dose (follow-up).
Population: The ADA evaluable set included all patients in the safety analysis set (i.e. those who had received any IP) who had non-missing baseline ADA data and at least 1 non-missing post-baseline ADA result.
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab | Durvalumab (MEDI4736) Monotherapy
Number analyzed (Participants) | 25 | 24
Participants
  ADA prevalence | 1 | 5
  ADA incidence | 0 | 3
  ADA pos post-baseline and pos at baseline | 0 | 0
  ADA pos post-baseline and not detected at baseline | 0 | 3
  ADA not detected post-baseline and pos at baseline | 1 | 2
  Treatment-boosted ADA | 0 | 0
  Persistent positive | 0 | 3
  Transient positive | 0 | 0
  Never positive | 24 | 19

11. Secondary Outcome: Presence of ADAs for Tremelimumab
Description: ADA prevalence was the proportion of the ADA evaluable set who had an ADA positive result at any point in time, baseline or post-baseline. ADA incidence (treatment-emergent ADA) was the sum of both treatment-induced (post-baseline ADA positive only) and treatment-boosted ADA positive patients as a proportion of the evaluable patient population. Treatment-boosted ADA was defined as baseline positive ADA titre boosted to a 4-fold or higher level following IP administration. Persistently positive was defined as positive at ≥2 post-baseline assessments (with ≥16 weeks between first and last positive) or positive at last post-baseline assessment. Transiently positive was defined as at least 1 post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive. Results are reported as number of patients with detectable anti- tremelimumab antibodies satisfying each of the indicated categories. Note: 'positive' is denoted by 'pos' in some category titles.
Time Frame: Immunogenicity samples were collected on Day 1 (Week 0), Week 4 and Week 12, and additionally at 3 months and 6 months after the last dose (follow-up).
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab
Number analyzed (Participants) | 25
Participants
  ADA prevalence | 2
  ADA incidence | 0
  ADA pos post-baseline and pos at baseline | 1
  ADA pos post-baseline and not detected at baseline | 0
  ADA not detected post-baseline and pos at baseline | 1
  Treatment-boosted ADA | 0
  Persistent positive | 0
  Transient positive | 1
  Never positive | 23

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event (TEAE) data is reported for the treatment period (up to 12 months) + follow-up (up to 90 days). Overall timeframe: up to approximately 15 months.
Description: TEAE definition: onset date ≥ first dose of IP (or pre-treatment AEs increasing in severity ≥ first dose) and ≤ the last dose of IP + 90 days or ≤ start date of subsequent therapy (whichever occurred first). All-cause mortality definition: death due to any cause (including disease progression of pancreatic cancer) up to 90 days after last dose of IP or until start of subsequent therapy, whichever occurred first.
Arm/Group | Durvalumab (MEDI4736) Plus Tremelimumab | Durvalumab (MEDI4736) Monotherapy
All-Cause Mortality (participants affected / at risk) | 19/32 | 16/32
Serious Adverse Events (participants affected / at risk) | 11/32 | 9/32
Other Adverse Events (participants affected / at risk) | 26/32 | 26/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (MEDI4736) Plus Tremelimumab (N=32) | Durvalumab (MEDI4736) Monotherapy (N=32)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) — Non-treatment related SAE in 1 patient with outcome equal to death.
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 2 (2)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 2 (3) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0) — Non-treatment related SAE in 1 patient with outcome equal to death
Infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) — Non-treatment related SAE in 1 patient with outcome equal to death
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 2 (2) — Non-treatment related SAE in 1 patient with outcome equal to death.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (MEDI4736) Plus Tremelimumab (N=32) | Durvalumab (MEDI4736) Monotherapy (N=32)
Hypothyroidism (Endocrine disorders) | 4 (4) | 0 (0)
Thyroiditis (Endocrine disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 5 (5) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 4 (6) | 5 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 6 (6) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (5) | 5 (6)
Vomiting (Gastrointestinal disorders) | 5 (6) | 5 (7)
Asthenia (General disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 6 (6) | 9 (10)
Feeling cold (General disorders) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 6 (10) | 2 (4)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Gingivitis (Infections and infestations) | 2 (2) | 2 (2)
Weight decreased (Investigations) | 2 (2) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 8 (9)
Hypophagia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (5) | 3 (6)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Study consisted of Part A Lead-in and 2 possible options for Part B: non-randomised expansion or randomised controlled trial. Criteria to open either option for Part B were not met and study was closed prematurely. Only Part A was conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-08-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT02558894/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT02558894/SAP_001.pdf